CLINICAL TRIAL: NCT00130884
Title: Effects of Peroral Levosimendan in the Prevention of Further Hospitalisations in Patients With Chronic Heart Failure. A Randomised, Phase II, Double-Blind, Placebo-Controlled, Multi-Centre, Parallel-Group Study
Brief Title: Peroral Levosimendan in Chronic Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3001081
Record Dates: First submitted 2005-08-15; First posted 2005-08-16 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2007-02

CONDITIONS: Chronic Heart Failure; Heart Diseases
Keywords: levosimendan; chronic heart failure; oral administration
MeSH Terms: conditions — Heart Diseases | interventions — Simendan

INTERVENTIONS:
Drug: levosimendan

SUMMARY:
The study will investigate the efficacy of oral levosimendan in patients with chronic New York Heart Association (NYHA) IIIb-IV heart failure (HF) using a composite end-point evaluating patient symptoms, morbidity and mortality. The patients are on treatment for at least 6 months.

DETAILED DESCRIPTION:
The patients are randomised to 3 groups; higher or lower levosimendan dose group or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed chronic heart failure
* Severe symptoms (NYHA IIIb-IV)
* Optimal on-going oral treatment for HF
* Left ventricular ejection fraction less than or equal to 30%

Exclusion Criteria:

* Severe obstruction of ventricular outflow tracts
* Acute myocardial infarction within 30 days before screening
* Cardiac surgery or coronary angioplasty within 30 days before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-03; Study Completion 2006-03

PRIMARY OUTCOMES:
Composite endpoint measuring symptoms, morbidity, mortality

CONTACTS AND LOCATIONS:
Overall Officials: Markku S Nieminen, MD, Principal Investigator — Helsinki University Central Hospital, Finland
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland